CLINICAL TRIAL: NCT03239977
Title: Social Intelligence Training for Custodial Grandmothers and Their Adolescent Grandchildren
Brief Title: Social Intelligence Training for Custodial Grandfamilies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kent State University (Other)
Responsible Party: Principal Investigator, Gregory Smith, Professor, Kent State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GCSmith RCT NIA
Record Dates: First submitted 2017-07-24; First posted 2017-08-04 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Emotional Intelligence; Quality of Life; Social Competence
Keywords: social intelligence; quality of life; social competence
MeSH Terms: conditions — Social Skills

STUDY DESIGN:
Intervention Model Description: Longitudinal Randomized Clinical Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Social Intelligence Training (Experimental): The Social Intelligence Intervention (SII) is delivered online to both custodial grandmothers and their adolescent grandchild separately. This is the sole active treatment condition within this RCT.
  Interventions: Behavioral: Online Social Intelligence Training
- Attention Control (AC) (Placebo Comparator): The attention control (AC) condition, known as The Healthy Living program provides information about different aspects of health.
  Interventions: Behavioral: Attention Control (AC)

INTERVENTIONS:
Behavioral: Online Social Intelligence Training — The SII consists of short 5-10 minute sessions organized into 7 modules designed to raise awareness of human nature and social relationships. The approach is based on evidence that SII is best advanced through interventions that modify key social cognitions regarding social engagement and enhance efficacy expectations regarding performance in social situations.
  Arms: Online Social Intelligence Training
Behavioral: Attention Control (AC) — A placebo condition delivered online to both custodial grandmothers and their adolescent grandchild which presents health-related information only.
  Arms: Attention Control (AC)

SUMMARY:
This study is a randomized clinical trial designed to compare an online social intelligence intervention with an active control condition at improving the emotional, physical, and social well-being of custodial grandmothers and their adolescent grandchildren,

DETAILED DESCRIPTION:
The investigators examine the efficacy of an online Social Intelligence Intervention (SII) at improving the health and well-being of custodial grandmothers (CGMs) and their adolescent custodial grandchildren (ACG) through mutual enhancement of their social competencies. This target population is of particular importance because both CGMs and ACG experience significant early life adversities that lead to hypervigilance of others, mistrust, social isolation, interpersonal conflict, and the inability to garner warmth and support from family and friends. Numerous studies have shown that these relational challenges within "risky families" often lead to life-long interpersonal difficulties that increase the probability of behavioral and physical health problems. Furthermore, adolescence is a key period for the development of social competence, which is influenced by supportive caregiving and positive modeling from female parent figures. However, because the ability of CGMs to carry out this intergenerational transmission of social skills is challenged, examining joint social intelligence training for CGM-ACG dyads is valuable for reversing this negative sequela. Yet, to date, no other investigators have done so. To address this gap, ant an online randomized clinical trial will be conducted with 340 nationally-recruited CGM-ACG (ages 12-18) dyads assigned to either the SII or an attention control condition. Data will be obtained at pre- and post-test, and at 3-, 6-, and 9-month follow-ups via questionnaires completed by phone. Daily dairies will be collected online from 170 randomly selected dyads, and qualitative interviews will be conducted with 60 dyads to probe how the SII affected their daily social competence and social ties. We will obtain quantitative and qualitative measures of key social cognitive processes, quality of close interpersonal ties, psychological well-being, and physical health. Administrative medical, criminal, and education records for all 340 dyads will also be obtained for cost-benefit analyses that examine changes in burden on public systems. These mixed-methods allow rigorous examination of four specific aims: (1) To investigate if the SII enhances social competencies that, in turn, produce long-term changes in relationship quality, well-being, and physical health; this includes determining if increased social competence in one dyad member leads to partner effects in the other; (2) To examine if cumulative risk, gender, and age moderate SII efficacy; (3) To study qualitatively how CGM-ACG dyads view the SII as having changed their social competencies and yielded positive outcomes; and (4) To assess the financial benefits of the SII to participants and their communities. These aims address a highly significant public health problem that will inform future efforts to support a wide range of high risk families, like custodial grandfamilies, who typically have insufficient access to formal support services. This SII is advantageous because it is inexpensive, delivered online, non-stigmatizing, and capable of reaching a target population that is geographically disperse and greatly in need of supportive programming.

ELIGIBILITY:
Inclusion Criteria:

* Grandmothers of any age or race
* Providing full-time care to an adolescent grandchild between ages 12-18
* Providing care in their own residence
* Providing care in total absence of the grandchild's biological parents.
* The target adolescent custodial grandchild will be of either gender
* Between ages 12- 18
* The custodial grandmother has provided full-time care for at least 6 months in total absence of the biological parents.
* Understanding of English well enough to comprehend all study materials.

Exclusion Criteria:

* Cognitive or behavioral problems that limit the ability of grandmothers and grandchildren to comprehend the intervention and complete study measures

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Grandmothers only will be eligible to participate
Enrollment: 680 (Estimated)
Dates: Start 2018-05-31 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Composite Latent Construct "Social Sensitivity" | Change will be assessed from baseline immediately post intervention, as well as at 3, 6, and 9 months post intervention.
  Measured by four standardized instruments self-report scales and daily diary entries
Change in Composite Latent Construct "Openness to Others" | Change will be assessed from baseline immediately post intervention, as well as at 3, 6, and 9 months post intervention
  Measured by two standardized self-report scales
Change in Composite Latent Construct "Social Self-Confidence" | Change will be assessed from baseline immediately post intervention, as well as at 3, 6, and 9 months post intervention
  Measured by three standardized self-report instruments
Change in Composite Latent Construct "Relationships and Social Ties" | Change will be assessed from baseline immediately post intervention, as well as at 3, 6, and 9 months post intervention
  Measures of ambivalence, close relationships, positive family connections, relationships with important groups; and social connections with peers.
Change in Physical Health | Change will be assessed from baseline immediately post intervention, as well as at 3, 6, and 9 months post intervention
  Self-reported health status measured by the Sf-12 Survey
Change in Composite Latent Construct "Psychological and Emotional Well-Being" | Change will be assessed from baseline immediately post intervention, as well as at 3, 6, and 9 months post intervention
  Separate measures of self-esteem, loneliness, depression, anxiety, introversion-extroversion, affective reactivity, social resilience

OTHER OUTCOMES:
Open Ended Interviews | Within one month after completing the social intelligence intervention.
  To be created open-ended measure of treatment satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Gregory C Smith, EdD, Principal Investigator — Kent State University
Locations (1):
- Kent State University, Kent, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Infurna FJ, Castro SA, Webster BA, Dolbin-MacNab ML, Smith GC, Crowley DM, Musil C. Does Social Intelligence Training Improve Daily Well-Being and Responsiveness to Daily Negative and Positive Events in Custodial Grandmothers? J Gerontol B Psychol Sci Soc Sci. 2024 Jul 1;79(7):gbae069. doi: 10.1093/geronb/gbae069. PMID 38695191
- [Derived] Smith GC, Infurna FJ, Dolbin-MacNab M, Webster B, Castro S, Crowley DM, Musil C, Hu L, Hancock GR. A Randomized Clinical Trial of Online Social Intelligence Training With Custodial Grandmothers. Gerontologist. 2024 May 1;64(5):gnad079. doi: 10.1093/geront/gnad079. PMID 37354201